CLINICAL TRIAL: NCT07302607
Title: Predictive Factors of Complete Response to Immunotherapy in Metastatic Melanoma: a Single-center Retrospective Study Between 2013 and 2021
Acronym: IMM
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9453
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Stage III Melanoma
Keywords: Stage III Melanoma; Immunotherapy in Metastatic Melanoma; Metastatic melanoma (unresectable stage III and IV)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although impressive progress has been made with this new therapeutic strategy, only a proportion of patients achieve a complete and sustained response. Studies have already identified predictive factors of treatment response that are now widely recognized. In this study, the investigators aim to identify other response factors not yet evaluated in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Unresectable stage III or stage IV melanoma according to the AJCC classification - 8th edition;
* Curative immunotherapy treatment (anti-PD-1 and/or anti-CTLA-4);
* Treatment and follow-up at the Dermatology Department of the Strasbourg University Hospitals;
* Immunotherapy initiated between January 1, 2013, and December 31, 2021.

Exclusion Criteria:

* Primary choroidal melanoma;
* Adjuvant-intent immunotherapy;
* Less than 3 months of follow-up after the start of immunotherapy;
* Change of treatment before the first reassessment;
* Treatment and follow-up at a department other than the Dermatology Department of the Strasbourg University Hospitals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject with unresectable stage III or stage IV melanoma according to the AJCC classification - 8th edition;
Sampling Method: Non-Probability Sample
Enrollment: 221 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors | 1 hour after consultation
  Response criteria
  Based on assessment of target and non-target lesions, the disease can be classified as 8:
  complete response (CR):
  requires all of:
  disappearance of all target and non-target lesions
  pathological lymph nodes must have reduced to <10 mm in short axis
  no new lesions
  partial response (PR):
  requires all of:
  at least 30% decrease in SOD of target lesions compared to baseline sum diameters (BSD)
  non-progressive disease of non-target lesions
  no new lesions
  progressive disease (PD):
  either one of:
  any new lesions
  at least 20% relative and 5 mm absolute increase of SOD of target lesions compared to smallest SOD ever recorded for the patient
  stable disease (SD):
  not meeting criteria for PD or PR

CONTACTS AND LOCATIONS:
Locations (1):
- Service de dermatologie - Réanimation - CHU de Strasbourg - France, Strasbourg, France